CLINICAL TRIAL: NCT03622346
Title: Periprosthetic Pathologic Fracture Following Tibial Echinococcosis: A Case Report
Brief Title: Periprosthetic Fracture Following Tibial Echinococcosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Hospitalar do Medio Tejo (Other)
Responsible Party: Principal Investigator, Germano Pereira Nascimento, Dr. Germano Nascimento, Principal Investigator, Centro Hospitalar do Medio Tejo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Echinococus treatment
Record Dates: First submitted 2018-07-19; First posted 2018-08-09 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Cystic Echinococcus
Keywords: Echinococcosis, Hydatidosis, TKR, Fracture
MeSH Terms: conditions — Echinococcosis; Fractures, Bone

STUDY DESIGN:
Intervention Model Description: Just one patient, subject to two surgeries: curettage and external fixation; subsequently the patient underwent total knee arthroplasty
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Semi-constrained total knee arthroplasty — Semi-constrained total knee arthroplasty

SUMMARY:
Cystic Echinococcus in the bone is rare, comprising 0.5% to 2.5% of all human hydatidosis Association of Hydatid disease to pathologic fractures involving knee prosthesis have not yet been described A combined surgical and medical approach is of paramount importance to avoid recurrence Resulting osseus defects is challenging and require specific prosthesis when treating this entity.

DETAILED DESCRIPTION:
Hydatid disease in humans caused by the parasitic tapeworm Echinococcus granulosus has an osseous involvement of about 0.5% to 2.5% of all cases in humans. The location of hydatid cysts in the tibia is seldom described in the medical literature, and its diagnosis and treatment is challenging.

This paper presents a patient, with a long term, well tolerated, bilateral total knee arthroplasty (TKA), treated at our clinic, with a recent history of pain and oedema in her left upper leg. After achieving a, radiologically and histopathologically, well documented, diagnosis of Echinococcosis lesion in her left proximal tibia, a surgical intervention was planed, a wide resection of the cyst performed, and a specific anti-helmintic therapy was instituted. Four years later the patient returns to the investigators observation complaining of pain and unable to bear weight on her left knee, from which a pathologic fracture, adjacent to the tibial component was diagnosed.

After surgical debridement of the newly advanced hydatid cyst growth, the TKA was revised, and due to the tibial component failure and the femoral implant loosening, a semi-constrained total knee revision arthroplasty was executed. Functional outcome was excellent.

Although challenges in treatment of musculoskeletal hydatid cysts (HC) lesions have been documented, data regarding the musculoskeletal HC lesions resembling tumor is scarce, and those resulting in a prosthetic failure haven't been published. The authors intend to add data concerning the therapeutic approach to this entity.

ELIGIBILITY:
Inclusion criteria

* Patients with echinococcus infection
* Patients which this infection compromises knee stability.

Exclusion criteria

* bacterial infection
* immunocompromised patients

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-01-05 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Pain assessed by numerical rating scale (NRS) | 6 years
  measured with numerical rating scale (NRS), ranging from 0 to 10 (minimum to maximum pain)

CONTACTS AND LOCATIONS:
Overall Officials: Germano P Nascimento, MD, Principal Investigator — Centro Hospitalar do Médio Tejo, EPE

IPD SHARING:
Plan to Share IPD: No
No personal patient information is to be made available.